CLINICAL TRIAL: NCT01420874
Title: Treatment of Advanced Colorectal or Pancreatic Cancer With Anti-CD3 x Anti-EGFR-Armed Activated T-Cells (Phase Ib)
Brief Title: Anti-CD3 x Anti-Erbitux® Armed Activated T Cells (Phase Ib) for Gastrointestinal (GI Cancer)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-025
Record Dates: First submitted 2011-08-17; First posted 2011-08-22 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Cancer of Pancreas; Pancreatic Neoplasm; Malignant Neoplasm of Large Intestine; Malignant Tumor of Colon; Colon Carcinoma; Cancer of Colon; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms | interventions — Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOX6 & EGFRBi armed ATC Infusions (Experimental): FOLFOX6: IV administration of 85 mb/m(2) oxaliplatin and 400 mg/m(2) leucovorin over 120 mins, followed by 400 mg/m(2) 5-fluorouracil (FU) bolus then 2400 mg/m(2) 5-FU as a 46 hr infusion. All patients must have central intravenous acess (e.g. mediport, PICC line) for continuous infusion of 5-FU. Adv. colorectal and pancreatic pts. w/no other standard chemo available, & in pts who cannot receive FOLFOX chemo, immunotherapy may be given w/o antecedent chemo.
  EGFRBi armed ATC Infusions: Armed ATC will be infused intravenously (IV) with the rate of infusion based on the endotoxin content of the product. All patients will be observed for at least 4 hours after an infusion. Armed ATC infusions will begin 3 weeks after chemotherapy and subsequent doses will be administered once weekly, for 3 weeks, then 12 weeks post aATC#1. Dose escalation level(per infusion): Level 0-5 billion; Level 1-10 billion; Level 2-20 billion; Level 3-40 billion
  Interventions: Drug: FOLFOX6; Biological: EGFRBi armed ATC Infusions

INTERVENTIONS:
Drug: FOLFOX6 — IV administration of 85 mb/m(2) oxaliplatin and 400 mg/m(2) leucovorin over 120 mins, followed by 400 mg/m(2) 5-fluorouracil (FU) bolus then 2400 mg/m(2) 5-FU as a 46 hr infusion. All patients must have central intravenous acess (e.g. mediport, PICC line) for continuous infusion of 5-FU. Adv. colorectal and pancreatic pts. w/no other standard chemo available, & in pts who cannot receive FOLFOX chemo, immunotherapy may be given w/o antecedent chemo.
  Other Names: leucovorin (FOLinic acid); Fluorouracil; OXaliplatin
Biological: EGFRBi armed ATC Infusions — Armed ATC will be infused intravenously (IV) with the rate of infusion based on the endotoxin content of the product. All patients will be observed for at least 4 hours after an infusion. Armed ATC infusions will begin 3 weeks after chemotherapy and subsequent doses will be administered once weekly, for 3 weeks, then 12 weeks post aATC#1. Dose escalation level(per infusion): Level 0-5 billion; Level 1-10 billion; Level 2-20 billion; Level 3-40 billion

SUMMARY:
The purpose of this research study is for the participant to give their own T cells (a type of blood cell in the body that can fight infections and possibly cancer) to them after they have been removed, grown in a lab, and then coated with an experimental drug.

This study will determine the highest dose of EGFR2Bi coated T cells that can be given without causing severe side effects. Initially a group of 3 participants will receive the same dose of study drug. If no serious side effects occur, the next group of participants will receive a slightly higher dose of study agent. The following groups of participants will receive higher doses of the study drug until a dose is reached where there are unacceptable side effects and maximum tolerated dose is found, or the planned highest dose level is reached with no side effects.

DETAILED DESCRIPTION:
The purpose of this study is to determine in a dose-escalation phase Ib trial the safety of 3 infusions of EGFR2Bi armed activated T cells (aATC), after chemotherapy, for patients with advanced colorectal and pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of colorectal or pancreatic adenocarcinoma
* Must have metastatic colorectal cancer or pancreatic cancer with stable disease after first line chemotherapy or patients with colorectal or pancreatic cancer who have progressed with standard chemotherapy options*
* Standard chemotherapy for metastatic colorectal cancer include 5-FU/capecitabine with either oxaliplatin or irinotecan based regimen with or without bevacizumab or cetuximab.
* Standard chemotherapy for metastatic pancreatic cancer include gemzar based regimen or FOLFIRINOX (5-FU, oxaliplatin, and irinotecan)
* Prior cetuximab, panitumumab, or other monoclonal antibody therapy allowed if given 28 days prior to the 1st infusion of armed T cells
* Absolute Neutrophil Count (ANC) ≥ 1,000/mm3
* Lymphocyte count ≥ 400/mm3
* Platelet Count ≥ 50,000/mm3
* Hemoglobin ≥ 8 g/dL
* Serum Creatinine < 2.0 mg/dl, Creatinine Clearance ≥50 ml/mm (can be calculated)
* Total Bilirubin ≤ 2 mg/dl (biliary stent is allowed)
* SGPT and SGOT < 5.0 times normal
* LVEF ≥ 45% at rest (MUGA or Echo)
* Pulse Oximetry of >88%
* Age ≥ 18 years at the time of consent
* Written informed consent and HIPAA authorization for release of personal health information
* Females of childbearing potential, and males, must be willing to use an effective method of contraception
* Females of childbearing potential must have a negative pregnancy test within 7 days of being registered for protocol therapy
* KPS ≥ 70% or SWOG Performance Status 0 or 1

Exclusion Criteria:

* Any chemotherapy related toxicities from prior treatment.(> grade I per CTCAE v4.0
* Known hypersensitivity to cetuximab or other EGFR antibody
* Treatment with any investigational agent within 14 days prior to being registered for protocol therapy Protocol version: 07/13/2011 8
* Symptomatic brain metastasis
* Chronic treatment with systemic steroids or another immuno-suppressive agent
* Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to being registered for protocol therapy
* Active liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* HIV infection
* Positive HbsAg
* Positive Hepatitis C
* Active bleeding or a pathological condition that is associated with a high risk of bleeding
* Uncontrolled systemic disease like active infections
* Nonmalignant medical illnesses that are uncontrolled or a controlled illness that may be jeopardized by the treatment with protocol therapy
* Females must not be breastfeeding
* Patient may be excluded if, in the opinion of the PI and investigator team, the patient is not capable of being compliant

Minor changes from these guidelines will be allowed at the discretion of the attending team under special circumstances. The reasons for exceptions will be documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08-17 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Determining in a dose-escalation phase Ib trial the safety of 3 infusions of EGFR2Bi aATC, and a booster infusion after 3 months, for patients with advanced colorectal or pancreatic cancer. | 4 wks after chemo, prior to ATC infusion #2; 1 wk later prior to ATC infusion #3; Wks 2, 4 & 9 post ATC infusion #3; Wk 8 post ATC #4 (booster)
  Participants will be assessed for changes in lab values (CBC, Sodium, potassium, calcium, magnesium, chloride, bicarbonate, glucose,BUN, creatinine, total Protein, albumin, total bilirubin, ALP, AST,ALT, CEA or CA 19-9.

SECONDARY OUTCOMES:
Determining whether IMT enhances anti-tumor immunity;Cytokine resp., phenotypic markers, anti-tumor cytotoxicity, in vivo and in vitro specific anti-tumor antibody prod. & molecular signaling markers of T-cell activation assessed before chemo & after IMT | 3 weeks after chemo prior to ATC infusion #1; At wks 4(ATC #2) & 5 (ATC #3) post chemo; wks 2 , 4 & 9 post ATC #3 infusion; Day of ATC #4 (booster infusion), then wks 2, 4 & 8; & mon 6 and 1yr post ATC #4 (booster infusion)
  Immune studies: Serum cytokine responses will be quantified focus on the levels of those factors known to be important regulators of T cell responses. Phenotype analysis will measure the percent of T, B, NKT and NK cells in peripheral blood mononuclear cell (PBMC) and tumor-infiltrating lymphocyte (TIL) samples. T cell proportions would be further analyzed by subset (CD4, CD8, CD25+). Cytotoxicity is measured in percentage in PBMC.
Determining the tumor response rate | Approximately every 8 weeks to until 1 year
  CT or PET Scan
Overall Survival | Approximately every 8 weeks to until 1 year
  CT or PET Scan

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Shields, M.D. PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Lum LG, Thakur A, Choi M, Deol A, Kondadasula V, Schalk D, Fields K, Dufrense M, Philip P, Dyson G, Aon HD, Shields AF. Clinical and immune responses to anti-CD3 x anti-EGFR bispecific antibody armed activated T cells (EGFR BATs) in pancreatic cancer patients. Oncoimmunology. 2020 Jun 10;9(1):1773201. doi: 10.1080/2162402X.2020.1773201. PMID 32939319